CLINICAL TRIAL: NCT04213885
Title: Safety and Effectiveness of the PXL Platinum 330 System for Corneal Collagen Cross-Linking With Corneal Thinning Conditions
Brief Title: Safety and Effectiveness of the PXL Platinum 330 System for Corneal Collagen Cross-Linking in Eyes With Corneal Thinning Position
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eye Specialists of Indiana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PXL330-001
Record Dates: First submitted 2019-12-27; First posted 2019-12-30 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Keratoconus, Unstable; Ectasia Corneal; Bacterial Keratitis
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin

STUDY DESIGN:
Intervention Model Description: Treatment of patients with disease
Who Masked: Outcomes Assessor
Masking Description: Randomized at outset
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pulsed Accelerated (Experimental): 30mW, 5 sec, 5 sec off, 10 minutes of illumination. Combination Product: PXL-330 Platinum device for cross linking with Peschke riboflavin solution will be used to load the cornea followed by UV-A cross linking of the cornea
  Interventions: Combination Product: PXL 330 Platinum device/Riboflavin
- Conventional (Active Comparator): 9mW continuous, 10 minutes of illumination. Combination Product: PXL-330 Platinum device for cross linking with Peschke riboflavin solution will be used to load the cornea followed by UV-A cross linking of the cornea
  Interventions: Combination Product: PXL 330 Platinum device/Riboflavin

INTERVENTIONS:
Combination Product: PXL 330 Platinum device/Riboflavin — 30mW, 5 sec, 5 sec off, 10 minutes of illumination

SUMMARY:
To determine whether the Peschke PXL-330 is safe and effective in the treatment of corneal thinning conditions.

DETAILED DESCRIPTION:
Patients with progressive keratoconus, pellucid marginal degeneration, infectious keratitis, or at risk for post-refractive corneal ectasia will be recruited and undergo epithelial-on corneal crosslinking with the Peschke PXL-330 system using pulsed, accelerated energy delivery. Patients will undergo monitoring for 1 year, with serial measurements of corneal topography, visual acuity, intraocular pressure and visual function questionnaire.

ELIGIBILITY:
Inclusion Criteria:Criterion 1,2,3 are required for all participants. Participants must also meet one or more of criteria 4-12. Criteria 13 is only relevant for contact lens wearers.

1. 12 years of age or older
2. Signed written informed consent
3. Willingness and ability to comply with schedule for follow-up visits
4. Presence of central or inferior steepening
5. Axial topography consistent with keratoconus, post-surgical ectasia, or pellucid marginal degeneration
6. Presence of one or more findings associated with keratoconus or pellucid marginal degeneration, such as

   1. Fleisher ring
   2. Vogt's striae
   3. Decentered corneal apex
   4. Munson's sign
   5. Rizzutti's sign
   6. Apical corneal scarring consistent with Bowman's breaks
   7. Scissoring of the retinoscopic reflex
   8. Crab-claw appearance on topography
7. Steepest keratometry (Kmax) value greater than or equal to 47.2
8. I-S keratometry difference < 1.5 D on the Pentacam map or topography map
9. Posterior corneal elevation > 16 microns
10. Thinnest corneal point <485 microns
11. Predicted Post LASIK/PRK stromal ablation depth <350 microns or expected keratometry >47.2, or patients undergoing PRK/SMILE in keratoconus suspect eyes
12. Bacterial or fungal keratitis persistent and not responding despite > 2 weeks of standard antimicrobial therapy or with rapid progression of corneal thinning, with loss of >25% corneal thickness
13. Contact lens wearers only:

    1. Removal of contact lenses for the require period of time prior to the screening refraction:

Contact Lens Type Discontinuations Time: Soft, 1 week; Soft Extended Wear, 2 weeks; Soft Toric, 3 weeks; Rigid Gas Permeable, 2 weeks per decade of wear -

Exclusion Criteria:

1. Eyes classified as normal or atypical normal on the severity grading scheme
2. Corneal pachymetry at the screening exam that is <300 microns at the the thinnest point in the eye(s) to be treated.
3. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example:

   1. History of or active corneal disease (e.g. herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, acanthamoeba, etc.)
   2. Clinically significant corneal scarring the CXL treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the cross-linking procedure.
4. Pregnancy (including plan to become pregnant) or lactation during the course of the study
5. A known sensitivity to the study medications
6. Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment of diagnostic tests.
7. Patients with a current condition that, in the physician's opinion, wold interfere with or prolong epithelial healing.

   -

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Mean keratometry in diopters | 1 year
  Average keratometry across the anterior topography of the cornea computed by a validated Scheimpflug topographer

SECONDARY OUTCOMES:
Best corrected visual acuity | 1 year
  Measurement of best corrected visual acuity on the validated early-treatment diabetic retinopathy study scale

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Specialists of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No